CLINICAL TRIAL: NCT07195370
Title: Evaluation of the Effectiveness of YAG Laser Iridotomy in Patients With Primary Angle-Closure: Temporal Peripheral Iridotomy Compared to Inferior Peripheral Iridotomy
Brief Title: Testing YAG Laser Iridotomy for Primary Angle-Closure Glaucoma
Acronym: yag laser PI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Afsaneh Naderi Beni, IsfahanUMS, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: feiz-123456; IR.MUI.MED.REC.1401.153 (Other: University of Isfahan Ethics Committee ID Issuing Organization)
Record Dates: First submitted 2025-08-26; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma Eye; Angle Closure Glaucoma
Keywords: Primary Angle-Closure Glaucoma
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Description: YAG laser peripheral iridotomy performed in the temporal region of one eye. Arm 2 Title (Other)
  Interventions: Other: peripheral iridotomy

INTERVENTIONS:
Other: peripheral iridotomy — This procedure involves using a neodymium-doped yttrium aluminum garnet (YAG) laser to create a small hole in the temporal region of the iris in one eye. It aims to relieve intraocular pressure in patients with primary angle-closure glaucoma by improving the flow of aqueous humor. The procedure is performed under local anesthesia in a clinical setting, with patients unaware of which eye receives this treatment. Outcomes, including laser power, intraocular pressure, visual symptoms, and complications, are monitored over six months.

SUMMARY:
This study evaluates the effectiveness and safety of YAG laser peripheral iridotomy performed at two different locations (temporal and inferior) in patients with primary angle-closure glaucoma, a leading cause of blindness worldwide. Patients visiting the glaucoma clinic at Feiz Hospital who are candidates for peripheral iridotomy will participate. In each patient, one eye will receive a temporal iridotomy, and the other eye will receive an inferior iridotomy, with patients unaware of the location used in each eye. The study will measure outcomes such as laser power, intraocular pressure, visual symptoms, and complications over six months to determine which approach is more effective and safer.

ELIGIBILITY:
Inclusion Criteria:Diagnosis of Primary Angle-Closure Glaucoma.

Adults (typically over 40 years old).

Ability to provide informed consent.

Narrow or closed anterior chamber angle (based on gonioscopy).

Intraocular pressure (IOP) controlled with medication but requiring surgery.

No previous iridotomy.

Exclusion Criteria:econdary glaucoma.

Active eye diseases (e.g., infection or inflammation).

Advanced cataracts or lens-related issues.

Severe visual impairment (e.g., less than 20/200 vision).

Uncontrolled systemic diseases (e.g., diabetes or cardiovascular disease).

Pregnancy or breastfeeding.

Previous eye surgery (except for minor procedures).

Inability to follow-up with scheduled visits.

-

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
adverse events | 1 day, 1 week, 1month
  Surgical and postoperative complications (e.g., bleeding, infection, or changes in intraocular pressure).

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No